CLINICAL TRIAL: NCT02221531
Title: Double-blind Randomised Non-inferiority Trial to Assess Efficacy and Safety of Carbetocin After Caesarean Section Applied as Iv-bolus as Compared to a Short-infusion
Brief Title: Carbetocin Trial: Carbetocin Appropriate Rate Better Equilibrium Between Tonus (TOnus) and CIrculatioN
Acronym: CARBETOCIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Obstetric Anaesthetists' Association United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-088
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Complications; Cesarean Section; Anesthesia; Reaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short infusion (Experimental): Carbetocin 100 microgram will be applied intravenously in a short infusion over about a minute
  Interventions: Drug: Carbetocin Short-infusion
- Bolus application (Other): Carbetocin 100 microgram will be applied intravenously by bolus application over about 15 seconds
  Interventions: Drug: Carbetocin Bolus application

INTERVENTIONS:
Drug: Carbetocin Short-infusion — Short-infusion of Carbetocin 100 microgram as compared to bolus application of Carbetocin 100 microgram (double dummy method)
  Arms: Short infusion
Drug: Carbetocin Bolus application — Carbetocin 100 microgram given intravenously as a bolus application over about 15 seconds
  Arms: Bolus application

SUMMARY:
Postpartum haemorrhage (PPH) is an obstetric emergency and defined as a blood loss of ≥500ml after vaginal birth and ≥1000ml after caesarean section (CS) and/or the need for blood transfusion within 24 hours after delivery (World Health Organization, Recommendations for the Prevention of Postpartum Haemorrhage. 2007; Leduc et al., J Obstet Gynaecol Can, 2009). Since PPH is more common after caesarean deliveries than after vaginal births and the rate of CS is rising over time and will probably continue to rise, the incidence of PPH is expected to increase accordingly.

A meta-analysis has shown that routine administration of an oxytocic agent after caesarean delivery leads to a reduced blood loss and decreases the risk of PPH (Cotter et al., Cochrane Database Syst Rev, 2001). The two most commonly used oxytocic drugs after operative delivery are oxytocin and carbetocin, a synthetic oxytocin-analogue. Carbetocin has the advantage over oxytocin of having a longer half-life and therefore reducing the use of additional uterotonics. Based on the findings of reduced cardiovascular side-effects with a short-infusion as compared to a bolus injection found for oxytocin (Thomas et al., Br J Anaesth, 2007), our study hypothesis is that a slower administration rate of carbetocin minimises the cardiovascular side effects without compromising the uterine tone. Therefore, we aim to investigate a short infusion of carbetocin 100 mcg applied in 100ml sodium chlorid compared to a bolus application in women undergoing primary or secondary caesarean delivery. This prospective, double-blind, randomised controlled non-inferiority trial will take place at the University Hospital Basel, Switzerland. We hypothesize uterine contraction not to be inferior (primary efficacy endpoint) and the mean arterial pressure to be higher after a short-infusion than after a bolus administration (primary safety endpoint).

ELIGIBILITY:
Inclusion Criteria:

* healthy women
* singleton pregnancy
* caesarean section under regional anaesthesia
* older than 18 years
* written informed consent

Exclusion Criteria:

* emergency caesarean section
* secondary caesarean section due to fetal distress
* comorbidities (cardiovascular, kidney or liver disorder, epilepsy)
* obstetric diseases (hypertension, (pre-)eclampsia)
* uterine malformation (including uterine fibroids)
* bleeding disorder
* known hypersensitivity to carbetocin or oxytocin
* fetal malformation

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Maximal uterine tone | within the first 5 minutes after cord clamping
  Uterine tone is assessed by the obstetrician on a linear analogue scale from 0 to 100

SECONDARY OUTCOMES:
Mean arterial pressure | within first five minutes after cord clamping
  mean arterial pressure is measured by a non-invasive blood pressure cuff at the upper arm

CONTACTS AND LOCATIONS:
Overall Officials: Salome Dell-Kuster, MD, Principal Investigator — Department of Anaesthesiology, University Hospital Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Dell-Kuster S, Hoesli I, Lapaire O, Seeberger E, Steiner LA, Bucher HC, Girard T. Efficacy and safety of carbetocin given as an intravenous bolus compared with short infusion for Caesarean section - double-blind, double-dummy, randomized controlled non-inferiority trial. Br J Anaesth. 2017 May 1;118(5):772-780. doi: 10.1093/bja/aex034. PMID 28498927
- [Derived] Dell-Kuster S, Hoesli I, Lapaire O, Seeberger E, Steiner LA, Bucher HC, Girard T. Efficacy and safety of carbetocin applied as an intravenous bolus compared to as a short-infusion for caesarean section: study protocol for a randomised controlled trial. Trials. 2016 Mar 22;17:155. doi: 10.1186/s13063-016-1285-5. PMID 27004531